CLINICAL TRIAL: NCT06342947
Title: A Randomized, Double-Blind, Placebo-Controlled Phase 2a Study Evaluating the Safety, Efficacy, Pharmacokinetics, and Pharmacodynamics of ALG-055009 in Non-Cirrhotic Adults With Metabolic Dysfunction-Associated Steatohepatitis
Brief Title: ALG-055009 in Non-cirrhotic Adults With MASH (HERALD)
Acronym: HERALD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Aligos Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: ALG-055009-303
Record Dates: First submitted 2024-03-15; First posted 2024-04-02 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-02

CONDITIONS: NASH; MASH; Metabolic Dysfunction-Associated Steatohepatitis; Nonalcoholic Steatohepatitis
Keywords: NASH; MASH; Metabolic Dysfunction-Associated Steatohepatitis; Nonalcoholic Steatohepatitis; Liver; Fatty Liver Disease; Liver Disease; THR-B; THR B; THR-β; THR β
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Liver Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- ALG-055009 softgel capsule 0.3mg (Experimental): ALG-055009 softgel capsule 0.3mg Daily for 12 weeks
  Interventions: Drug: ALG-055009
- ALG-055009 softgel capsule 0.5mg (Experimental): ALG-055009 softgel capsule 0.5mg Daily for 12 weeks
  Interventions: Drug: ALG-055009
- ALG-055009 softgel capsule 0.7mg (Experimental): ALG-055009 softgel capsule 0.7mg Daily for 12 weeks
  Interventions: Drug: ALG-055009
- ALG-055009 softgel capsule 0.9mg (Experimental): ALG-055009 softgel capsule 0.9mg Daily for 12 weeks
  Interventions: Drug: ALG-055009
- Placebo (Placebo Comparator): Placebo softgel capsule Daily for 12 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ALG-055009 — Softgel Capsule
  Arms: ALG-055009 softgel capsule 0.3mg; ALG-055009 softgel capsule 0.5mg; ALG-055009 softgel capsule 0.7mg; ALG-055009 softgel capsule 0.9mg
Drug: Placebo — Softgel Capsule
  Arms: Placebo

SUMMARY:
This is a Phase 2a study to evaluate the safety, tolerability, efficacy, pharmacokinetics, and pharmacodynamics of oral (PO) daily (QD) doses of ALG-055009 (soft gelatin [softgel] capsule) for 12 weeks.

DETAILED DESCRIPTION:
This is a double-blind, randomized, placebo-controlled Phase 2a study to evaluate the safety, tolerability, efficacy, pharmacokinetics, and pharmacodynamics of oral (PO) daily (QD) doses of ALG-055009 (soft gelatin [softgel] capsule) for 12 weeks. The study will be conducted in approximately 100 adult non-cirrhotic subjects with presumed MASH and liver fibrosis (F1-F3). The study will be conducted at up to approximately 45 sites throughout the United States of America.

ELIGIBILITY:
Key Inclusion Criteria:

* Male or female, 18 to 75 years of age
* Body mass index (BMI) ≥ 25 kg/m2
* Diagnosis of presumed NASH/MASH with F1-F3 liver fibrosis based on one of the following:

  * Liver biopsy within 6 months prior to screening showing a NAFLD activity score (NAS) of ≥4 with at least a score of 1 in each of the NAS components; OR
  * Having ≥2 metabolic syndrome criteria and a screening FibroScan liver stiffness measurement between 7 - 20 kPa
* Screening FibroScan with CAP score of >300 dB/m
* Screening MRI-PDFF with ≥10% liver fat content

Key Exclusion Criteria:

* History or clinical evidence of chronic liver disease other than metabolic dysfunction-associated steatotic liver disease (MASLD)
* History or current evidence of cirrhosis
* History of liver transplantation or known planned liver transplantation
* History or current evidence of a pituitary disorder or hyperthyroidism
* Untreated clinical or subclinical hypothyroidism; or on thyroid replacement therapy at screening or within the last 6 months prior to screening.
* TSH, free T4, or Total T3 >1.1 x ULN or <0.9 x LLN
* Clinically concerning abnormal ECG or cardiac history
* HbA1c ≥9.5%
* Platelet count ≤135,000/mm3
* ALT or AST >5 x ULN
* INR >1.3
* Albumin <3.5 g/dL
* eGFR <45 mL/min/1.73 m2

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2024-08-19 (Actual); Study Completion 2024-09-09 (Actual)

PRIMARY OUTCOMES:
Percent relative change from baseline in liver fat content | 12 weeks
  Percent relative change from baseline in liver fat content by MRI-PDFF at Week 12

SECONDARY OUTCOMES:
Absolute change from baseline in liver fat content | 12 weeks
  Absolute change from baseline in liver fat content by MRI-PDFF at Week 12
Proportion of subjects with ≥30% relative reduction in liver fat content | 12 weeks
  Proportion of subjects with ≥30% relative reduction in liver fat content by MRI-PDFF at Week 12
Proportion of subjects with ≥50% relative reduction in liver fat content | 12 weeks
  Proportion of subjects with ≥50% relative reduction in liver fat content by MRI-PDFF at Week 12
Proportion of subjects with ≥70% relative reduction in liver fat content | 12 weeks
  Proportion of subjects with ≥70% relative reduction in liver fat content by MRI-PDFF at Week 12
Proportion of subjects with normalization (<5%) in liver fat content | 12 weeks
  Proportion of subjects with normalization (<5%) in liver fat content by MRI-PDFF at Week 12

OTHER OUTCOMES:
Change from baseline (absolute/percent) in lipid/lipoprotein levels | 12 weeks
  Change from baseline (absolute/percent) in lipid/lipoprotein levels at Week 12
Change from baseline (absolute/percent) in SHBG | up to 16 weeks
  Change from baseline (absolute/percent) in SHBG
Change from baseline (absolute/percent) alanine aminotransferase (ALT) | 12 weeks
  Change from baseline (absolute/percent) in alanine aminotransferase (ALT) at Week 12
Change from baseline (absolute/percent) aspartate aminotransferase (AST) | 12 weeks
  Change from baseline (absolute/percent) in aspartate aminotransferase (AST) at Week 12
Safety and tolerability will be assessed by monitoring TEAEs | 16 weeks
  Safety and tolerability will be assessed by monitoring TEAEs
Safety and tolerability will be assessed by monitoring 12-lead electrocardiograms (ECGs) | 16 weeks
  Safety and tolerability will be assessed by monitoring 12-lead electrocardiograms (ECGs)
PK parameters of ALG-055009 in plasma, AUCs | 12 weeks
  PK parameters of ALG-055009 in plasma, AUCs
PK parameters of ALG-055009 in plasma, Tmax | 12 weeks
  PK parameters of ALG-055009 in plasma, Tmax
PK parameters of ALG-055009 in plasma, Cmax | 12 weeks
  PK parameters of ALG-055009 in plasma, Cmax
PK parameters of ALG-055009 in plasma, Cmin | 12 weeks
  PK parameters of ALG-055009 in plasma, Cmin

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Harrison, MD, Principal Investigator
Locations (40):
- United States (40):
  - Aligos Clinical Study Site 18, Chandler, Arizona
  - Aligos Clinical Study Site 15, Peoria, Arizona
  - Aligos Clinical Study Site 17, Tucson, Arizona
  - Aligos Clinical Study Site 35, Chula Vista, California
  - Aligos Clinical Study Site 1, Lincoln, California
  - Aligos Clinical Study Site 37, Poway, California
  - Aligos Clinical Study Site 10, Rialto, California
  - Aligos Clinical Study Site 26, Bradenton, Florida
  - Aligos Clinical Study Site 25, Clearwater, Florida
  - Aligos Clinical Study Site 39, Fort Myers, Florida
  - Aligos Clinical Study Site 2, Maitland, Florida
  - Aligos Clinical Study Site 22, Ocoee, Florida
  - Aligos Clinical Study Site 32, Port Orange, Florida
  - Aligos Clinical Study Site 38, Sarasota, Florida
  - Aligos Clinical Study Site 31, The Villages, Florida
  - Aligos Clinical Study Site 3, Viera, Florida
  - Aligos Clinical Study Site 30, Winter Park, Florida
  - Aligos Clinical Study Site 23, Athens, Georgia
  - Aligos Clinical Study Site 12, Topeka, Kansas
  - Aligos Clinical Study Site 29, Louisville, Kentucky
  - Aligos Clinical Study Site 24, Bastrop, Louisiana
  - Aligos Clinical Study Site 5, Houma, Louisiana
  - Aligos Clinical Study Site 4, Marrero, Louisiana
  - Aligos Clinical Study Site 6, Metairie, Louisiana
  - Aligos Clinical Study Site 14, Chesterfield, Michigan
  - Aligos Clinical Study Site 7, New York, New York
  - Aligos Clinical Study Site 8, Morehead City, North Carolina
  - Aligos Clinical Study Site 21, Columbus, Ohio
  - Aligos Clinical Study Site 16, Westlake, Ohio
  - Aligos Clinical Study Site 36, East Greenwich, Rhode Island
  - Aligos Clinical Study Site 9, Nashville, Tennessee
  - Aligos Clinical Study Site 19, Austin, Texas
  - Aligos Clinical Study Site 33, Bellaire, Texas
  - Aligos Clinical Study Site 27, Brownsville, Texas
  - Aligos Clinical Study Site 28, Edinburg, Texas
  - Aligos Clinical Study Site 40, Farmers Branch, Texas
  - Aligos Clinical Study Site 20, San Antonio, Texas
  - Aligos Clinical Study Site 11, Waco, Texas
  - Aligos Clinical Study Site 13, Manassas, Virginia
  - Aligos Clinical Study Site 34, Seattle, Washington